CLINICAL TRIAL: NCT06390072
Title: The Impact of a Brief Hypnosis Intervention on Single-limb Dynamic Balance in People With Chronic Ankle Instability: Enhancing and Limiting Psychological Factors, Perceived and Performance-based Ankle Stability, and Heart-rate Variability
Brief Title: Project Hypnos: The Impact of a Brief Hypnosis Intervention on Single-limb Dynamic Balance in People With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-X-71
Record Dates: First submitted 2024-04-02; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Ankle Sprains; Motor Coordination or Function; Developmental Disorder
Keywords: Interoceptive awareness; Heart rate variability; Anxiety
MeSH Terms: conditions — Ankle Injuries; Developmental Disabilities; Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: This basic experimental pilot study involved a randomized cross-over design of two brief interventions with a 1:1 allocation ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-hypnosis (Experimental): The audio-guided self-hypnosis practice was sourced from the Reveri App (reveri.com), developed by Dr. David Spiegel, and entitled "Hypnosis Prep for Workout"
  Interventions: Behavioral: Self-Hypnosis; Behavioral: Ankle Education
- Ankle Education (Active Comparator): The ankle education video, entitled "Ankle Sprain Rehab Exercises" was sourced from the Physio Tutors YouTube channel
  Interventions: Behavioral: Self-Hypnosis; Behavioral: Ankle Education

INTERVENTIONS:
Behavioral: Self-Hypnosis — Participants listened to an 8-minute audio-guided self-hypnosis related to improving their physical performance
Behavioral: Ankle Education — Participants listened to an 8-minute video on ankle sprain diagnosis, prognosis, and treatment

SUMMARY:
This study will determine the relationship of one's self-reported awareness of their body and their ankle motor control for people with chronic ankle instability. This study will further identify the correlates between certain psychological characteristics (i.e., fear and anxiety) and autonomic nervous system arousal (i.e., heart rate variability). Furthermore, this study will elucidate the potential impact of a brief hypnosis practice on balance performance.

ELIGIBILITY:
Inclusion Criteria:

* History of one significant ankle sprain
* Experiences of instability in the ankle, determined by a score of > 11 on the Identification of Functional Ankle Instability (IdFAI) questionnaire
* An overall sensation of disability, determined by a score of < 90% on the Functional Ankle Ability Measure (FAAM) questionnaire

Exclusion Criteria:

* If the participant's initial ankle sprain was within the past twelve months or the most recent ankle sprain was within the past three months, the participant was excluded from eligibility
* A history of lower extremity surgery
* A fracture to the lower extremity
* Any acute musculoskeletal injuries to lower extremities in the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Balance test 1 | Through the study completion, up to 8 days from baseline assessment. Assessed at pre-intervention and post-intervention for sessions 1 and 2
  Biodex Stability System
Balance test 2 | Through the study completion, up to 8 days from baseline assessment. Assessed at pre-intervention and post-intervention for sessions 1 and 2
  Y-Balance test
Heart rate variability | Through the study completion, up to 8 days from baseline assessment. Assessed at pre-intervention and post-intervention for sessions 1 and 2
  HRV was captured for 5 minutes using a three-lead electrocardiogram at the beginning of each of the two lab sessions

SECONDARY OUTCOMES:
Ankle disability measure 1 | T0, Baseline/Enrollment
  Identification of Functional Ankle Instability, used for eligibility screening
Ankle disability measure 2 | T0, Baseline/Enrollment
  Functional Ankle Ability Measure
Interoceptive awareness measure 1 | T0, Baseline/Enrollment
  Mindful Presence - Bodily Awareness
Interoceptive awareness measure 2 | T0, Baseline/Enrollment
  Multidimensional Assessment of Interoceptive Awareness (MAIA-2)
Emotional Distress-Anxiety | T0, Baseline/Enrollment
  PROMIS Emotional Distress-Anxiety item bank
Kinesiophobia | T0, Baseline/Enrollment
  Tampa Scale of Kinesiophobia (TSK-11)
Pain self-efficacy | T0, Baseline/Enrollment
  Pain Self-Efficacy Questionnaire (PSEQ-10)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Karayannis, MPT, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided